CLINICAL TRIAL: NCT03661515
Title: An Investigator Sponsored Phase I Trial of Selinexor (KPT-330) Plus FLAG-Ida for the Treatment of Relapsing/Refractory AML
Brief Title: Selinexor (KPT-330) Plus FLAG-Ida for the Treatment of Relapsing/Refractory AML
Acronym: FLAGINEXOR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FLAGINEXOR: IST-ESP-000155
Record Dates: First submitted 2018-07-17; First posted 2018-09-07 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; Relapsed; Refractory; Selinexor
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence | interventions — selinexor; fludarabine; Idarubicin; Cytarabine; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fludarabine-Idarubicine-Cytarabine- Selinexor (Experimental): fludarabine 30 mg/m2/day intravenously on days 1 to 4, idarubicin 10 mg/m2/day intravenously on days 1 to 3, cytarabine 2 g/m2/day intravenously on days 1 to 4, G-CSF 300 mcg/m2/day subcutaneously from days -1 to 5. This schedule will be combined with oral selinexor (KPT-330) for three weeks at days and dose according to escalation level:
  * Level -1: Selinexor 40 mg/day, once weekly
  * Level 1: Selinexor 60 mg/day, once weekly
  * Level 2: Selinexor 80 mg/day, once weekly
  * Level 3: Selinexor 100 mg/day, once weekly
  Interventions: Drug: Selinexor; Drug: fludarabine; Drug: idarubicin; Drug: cytarabine; Drug: G-CSF

INTERVENTIONS:
Drug: Selinexor — According to escalation level:
  * Level -1: Selinexor 40 mg/day, once weekly
  * Level 1: Selinexor 60 mg/day, once weekly
  * Level 2: Selinexor 80 mg/day, once weekly
  * Level 3: Selinexor 100 mg/day, once weekly
Drug: fludarabine — fludarabine 30 mg/m2/day intravenously on days 1 to 4
Drug: idarubicin — idarubicin 10 mg/m2/day intravenously on days 1 to 3
Drug: cytarabine — cytarabine 2 g/m2/day intravenously on days 1 to 4
Drug: G-CSF — G-CSF 300 mcg/m2/day subcutaneously from days -1 to 5

SUMMARY:
This protocol corresponds to a multicenter, open-label, non-randomized, phase I study designed to determine the safety of the combination of selinexor with chemotherapy in young patients with relapsed or refractory AML.

The clinical trial is divided into pre-treatment, treatment (induction and consolidation cycles) and follow-up periods and consists of a phase I design in which es-calating doses of selinexor will be given to 3 groups, each with 3-6 patients until achieving the maximum tolerated dose (MTD).

DETAILED DESCRIPTION:
Study Design:

This protocol corresponds to a multicenter, open-label, non-randomized, phase I study designed to determine the safety of the combination of selinexor with chemotherapy in young patients with relapsed or refractory AML.

The clinical trial is divided into pre-treatment, treatment (induction and consolidation cycles) and follow-up periods and consists of a phase I design in which es-calating doses of selinexor will be given to 3 groups, each with 3-6 patients until achieving the maximum tolerated dose (MTD).

Each cycle (second induction, consolidation or maintenance) of treatment will compromise 3 weeks of selinexor treatment, and at least one week off treatment. The new cycle will not start if there is an ongoing grade 3 or higher non-hematologic toxicity or persistent grade 3 neutropenia in patients achieving CR.

Study design allows a maximum of 18 patients.

Induction cycle (up to 2 cycles):

Treatment will consist of fludarabine 30 mg/m2/day intravenously on days 1 to 4, idarubicin 10 mg/m2/day intravenously on days 1 to 3, cytarabine 2 g/m2/day intravenously on days 1 to 4, G-CSF 300 mcg/m2/day subcutaneously from days -1 to 5. This schedule will be combined with oral selinexor (KPT-330) for three weeks at days and dose according to escalation level:

* Level -1: Selinexor 40 mg/day, once weekly
* Level 1: Selinexor 60 mg/day, once weekly
* Level 2: Selinexor 80 mg/day, once weekly
* Level 3: Selinexor 100 mg/day, once weekly If a partial response is obtained after the first cycle of treatment, an identical induction therapy will be administered.

If a patient achieves a complete remission after 1 or 2 cycles of FLAG-IDA plus selinexor, allogeneic stem cell transplantation (Allo-SCT) will be attempted. If Allo-SCT is not possible, this patient will receive consolidation treatment as described below.

Consolidation cycle (up to 2 cycles):

Treatment will consist of cytarabine 1 g/m2/day intravenously (3 hours) on days 1 to 6. This schedule will be combined with oral selinexor (the same dosage that was administered to the patient in the induction cycle).

At most, patients will receive up to 4 cycles of combined chemotherapy.

Maintenance cycle:

For patients in CR, and when an Allo-SCT is not feasible, a maintenance treatment with selinexor could be started for up to 6 cycles.

Selinexor will be given at the same level as during induction therapy in cycles of four weeks (3 weeks on selinexor and 1 week off).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent in accordance with national, local, and institutional guidelines. The patient must provide informed consent prior to the first screening procedure.
* Age ≥ 18, and ≤ 65 years old.
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2.
* Diagnosis of AML (defined using WHO criteria) of any type except for acute promyelocytic leukemia (APL; AML M3).
* Relapsing or refractory AML, defined as either:

Recurrence of disease after first CR (duration of CR ≤ 24 months), or Failure to achieve CR or CRi after 1 or 2 identical induction cycles containing an anthracycline plus cytarabine based schedule.

* No contraindications to receive intensive chemotherapy.
* Female patients of child-bearing potential must have a negative serum pregnancy test at screening and agree to use two reliable methods of contraception for three months after their last dose of medication. Male patients must use a reliable method of contraception (if sexually active with a female of child-bearing potential).
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests and other study procedures.

Exclusion Criteria:

* Patients with APL/AML M3.
* Patients who are pregnant or lactating.
* Radiation, chemotherapy, or immunotherapy or any other anticancer therapy ≤ 2 weeks prior to Cycle 1 Day 1 or radio-immunotherapy 4 weeks prior to Cycle 1 Day 1. Hydroxyurea is permitted until 1 day prior to Cycle 1 Day 1.
* Previous treatment with a SINE compound.
* Major surgery within 2 weeks of first dose of study drug.
* Any life-threatening illness, medical condition or organ system dysfunction which, in the Investigator's opinion, could compromise the patient's safety.
* Unstable cardiovascular function:

  * Symptomatic ischemia, or uncontrolled clinically significant conduction abnormalities (i.e., ventricular tachycardia on anti-arrhythmia are excluded; 1st degree AV block or asymptomatic LAFB/RBBB will not be excluded), or congestive heart failure (CHF) of NYHA Class ≥ 3, or myocardial infarction (MI) within 3 months.
* Uncontrolled (i.e., clinically unstable) infection requiring parenteral antibiotics, antivirals, or antifungals within one week prior to first dose; however, prophylactic use of these agents is acceptable even if parenteral.
* Active hepatitis B or hepatitis C infection.
* Known human immunodeficiency virus (HIV) infection (HIV testing is not required as part of this study).
* Patients unable to swallow tablets, patients with malabsorption syndrome, or any other gastrointestinal (GI) disease or GI dysfunction that could interfere with absorption of study treatment.
* Any of the following laboratory abnormalities unless due to leukemia:

  * Hepatic dysfunction: bilirubin > 2.0 times the upper limit of normal (ULN) (except patients with Gilbert's syndrome: total bilirubin of > 3 x ULN) and alanine aminotransferase (ALT) and aspartic aminotransferase (AST) > 2.5 times ULN or in case of liver metastases: In patients with known liver involvement of their cancer, AST and ALT > 5 x ULN.
  * Severe renal dysfunction: estimated creatinine clearance of < 30 mL/min, measured in 24 hour urine or calculated using the formula of Cockroft and Gault: (140-Age) x Mass (kg)/[72 x creatinine (mg/dL)]; multiply by 0.85 if female

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-07-17 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of selinexor in combination with FLAG-Ida regimen | At the end of Cycle 1 (each cycle is 56 days)
  A standard 3 + 3 dose escalation schedule will be used for all escalations. Initially, three patients will be entered in each cohort at the scheduled starting dose level for that cohort. If a drug-related DLT (see Section 5.1.5.3) is not seen at the scheduled dose, the dose will be escalated for the subsequent group of 3 patients.
  If 1 of 3 patients experiences a drug-related DLT, then 3 additional patients will receive that dose. If ≤ 2 of 6 patients experiences a drug-related DLT, the next scheduled dose level will be available. If, at a given dose level, > 2 patients experience a drug-related DLT, the MTD will have been exceeded, additional enrollment within that cohort will cease, and dose escalation will stop.
  If a dose level proves intolerable (≥ 3 patients experience a DLT), enrollment will proceed at one dose-level lower.
Find recommended phase 2 dose | 3 months
  A standard 3 + 3 dose escalation schedule will be used for all escalations. Initially, three patients will be entered in each cohort at the scheduled starting dose level for that cohort. If a drug-related DLT (see Section 5.1.5.3) is not seen at the scheduled dose, the dose will be escalated for the subsequent group of 3 patients.
  If 1 of 3 patients experiences a drug-related DLT, then 3 additional patients will receive that dose. If ≤ 2 of 6 patients experiences a drug-related DLT, the next scheduled dose level will be available. If, at a given dose level, > 2 patients experience a drug-related DLT, the MTD will have been exceeded, additional enrollment within that cohort will cease, and dose escalation will stop.
  If a dose level proves intolerable (≥ 3 patients experience a DLT), enrollment will proceed at one dose-level lower.

SECONDARY OUTCOMES:
Assessment of toxicity: Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 1 year
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0.
CR and CRi | 3 months
  antileukemic effects, including its ability to produce complete remissions, of Selinexor in combination with chemotherapy

CONTACTS AND LOCATIONS:
Locations (4):
- Spain (4):
  - Hospital Germans Tries i Pujol, Badalona, Badalona
  - Hospital San Pedro de Alcántara,, Cáceres
  - Hospital Universitario 12 de Octubre,, Madrid
  - Hospital la Fe, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martinez Sanchez MP, Megias-Vericat JE, Rodriguez-Veiga R, Vives S, Bergua JM, Torrent A, Suarez-Varela S, Boluda B, Martinez-Lopez J, Cano-Ferri I, Acuna-Cruz E, Torres-Minana L, Martin-Herreros B, Serrano A, Sempere A, Barragan E, Sargas C, Sanz M, Martinez-Cuadron D, Montesinos P; PETHEMA group. A phase I trial of selinexor plus FLAG-Ida for the treatment of refractory/relapsed adult acute myeloid leukemia patients. Ann Hematol. 2021 Jun;100(6):1497-1508. doi: 10.1007/s00277-021-04542-8. Epub 2021 Apr 29. PMID 33914097